CLINICAL TRIAL: NCT05397275
Title: The Effect of Progressive Relaxation and Breathing Exercise on Sleep Quality and Exercise Self-Efficacy in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Kevser Sevgi Ünal Aslan, assistant professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: osmaniye korkut ata university
Record Dates: First submitted 2022-05-20; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: COPD Asthma
Keywords: Exercise Self-Regulatory Efficacy,; sleep quality; PGE with breathing exercises; pulmonary rehabilitation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): progressive muscle relaxation exercises + breathing exercise
  Interventions: Other: progressive muscle relaxation+breathe exercises
- control group (Experimental): only breathing exercise
  Interventions: Other: breathe exercises

INTERVENTIONS:
Other: progressive muscle relaxation+breathe exercises — progressive muscle relaxation+breathe exercises
  Arms: experimental group
Other: breathe exercises — breathe exercises
  Arms: control group

SUMMARY:
Aim: This study was conducted to determine the effect of progressive muscle relaxation and breathing exercise on sleep quality and exercise self-efficacy in chronic obstructive pulmonary patients.

Methods: This study was conducted as a randomized controlled experimental study. The study was conducted with 64 chronic obstructive pulmonary patients, where 36 of them were in the intervention group and 34 in the control group. Data of the study were collected using the descriptive information form, the Pittsburgh Sleep Quality Index, and the Exercise Self-Regulatory Efficacy Scale (Ex-SRES) for patients with COPD.

Results: When the total scores pertaining to the sleep quality index and exercise self-efficacy of the individuals in the intervention and control groups were compared, it was found that there were statistically significant differences in the intervention group compared to the control group (p < 0.05).

Keywords: Exercise Self-Regulatory Efficacy, sleep quality in patients with COPD, PGE along with breathing exercises, pulmonary rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* were to be 18 years of age or older
* not using sleeping pills
* verbally stating that they have moderate and severe sleep disorders.

Exclusion Criteria:

* having any lung disease other than COPD
* having cardiological problems (heart failure, uncontrollable hypertension, history of angina and myocardial infarction, heart valve problems), psychotic disorder,
* inability to communicate verbally and having hearing problems.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
progressive muscle relaxation exercises changes sleep quality and exercise self-efficacy. | 1 mounth
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index as an pre- test and 4 weeks later as a post-test test.

SECONDARY OUTCOMES:
progressive muscle relaxation exercises with breathing exercise changes sleep quality and exercise self-efficacy. | 1 mounth
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index as an pre-test and 4 weeks later as a post-test.
  .The Exercise Self-Regulatory Efficacy Scale will be used as a pre-test and after 4 weeks as a post-test to measure the exercise capacity of COPD patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
may be published at the discretion of the authors, provided appropriate justifications are provided.